CLINICAL TRIAL: NCT02231125
Title: Efficacy and Safety of Abelmoschus Manihot for IgA Nephropathy: a Multicentre, Double-blind, Double-dummy, Randomized Controlled Trial
Brief Title: Efficacy and Safety of Abelmoschus Manihot for IgA Nephropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Xiangmei (Other)
Collaborators: Jiangsu Suzhong Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Chen Xiangmei, professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S2014-039-01
Record Dates: First submitted 2014-08-30; First posted 2014-09-04 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: IgA Nephropathy
Keywords: Abelmoschus manihot; IgA Nephropathy; proteinuria; efficacy; safety
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria | interventions — Losartan; Huangkui

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abelmoschus manihot (AM) (Experimental): Abelmoschus manihot (AM): Huangkui capsule (Jiangsu Suzhong Pharmaceutical Group Co., Ltd.), 0.5 g × 30 capsules/box. A huangkui capsule is a single plant drug extract of Flos Abelmoschus manihot.
  Interventions: Drug: Abelmoschus manihot
- Losartan (Experimental): Losartan potassium (Hangzhou MSD Pharmaceutical Co., Ltd.), 100 mg × 7 capsules/box.
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — Losartan potassium tablet 100mg/time, once /day plus Huangkui Capsule dummy 2.5g/time, thrice /day, all drug and dummy are taken orally every day for 48 weeks during the whole study process.
  Other Names: Cozaar
  Arms: Losartan
Drug: Abelmoschus manihot — Huangkui Capsule 2.5g/time, thrice /day plus Losartan potassium tablet dummy 100mg/time, once /day, all drug and dummy are taken orally every day for 48 weeks during the whole study process.
  Other Names: Huangkui Capsule
  Arms: Abelmoschus manihot (AM)

SUMMARY:
-IgA nephropathy is the most common primary glomerular disease in China, Huangkui Capsule is a single medicament of traditional Chinese medicine consists of Abelmoschus manihot and has been widely used to treat kidney disease. The purpose of this study is to evaluate the safety and efficacy of Abelmoschus manihot for treating IgA nephropathy in large scale samples with long time take.

DETAILED DESCRIPTION:
The test has not been completed .

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosed as chronic nephritic syndrome
* IgA nephropathy diagnosed by kidney biopsy
* Aged from 18 to 65 years，male or female
* Blood pressure of ≤140/90mmHg
* Estimated Glomerular Filtration Rate (eGFR)≥45ml/min/1.73 m2
* 24-hour proteinuria ranged between 0.5g-3.0g
* Obtaining the signed informed consent from patients

Exclusion Criteria:

* Secondary IgA nephropathy
* Be allergic to Huangkui Capsule or Losartan potassium tablet
* Taken Huangkui Capsule or ACEI or ARB in last 6 weeks
* Taken the glucocorticoids, immunosuppressants or common threewingnut root and such as drugs with immunosuppressive actions in the last 12 months
* Blood pressure <90/60mmHg
* Serum potassium level > 5.5mmol / L
* Serum albumin level <30g / L
* Lactation, pregnancy or plans pregnancy during the study period
* Unilateral or bilateral renal artery stenosis
* Combined with severe primary diseases of heart, brain, liver and hematopoietic system and so on, or other serious diseases which can affect the patient's life
* Participating in another clinical study in the same period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in 24-h proteinuria from baseline after treatment | Baseline(week 0), week 4, week 12, week 24, week 36, week 48

SECONDARY OUTCOMES:
Change in serum creatinine from baseline after treatment | Baseline(week 0), week 4, week 12, week 24, week 36, week 48
Change in estimated glomerular filtration rate (eGFR) from baseline after treatment | Baseline(week 0), week 4, week 12, week 24, week 36, week 48

CONTACTS AND LOCATIONS:
Overall Officials: Xiangmei Chen, MD.& Ph.D, Principal Investigator — Department of Nephrology,State Key Laboratory of Kidney Disease,National Clinical Research Center for Kidney Disease, Chinese PLA General Hospital
Locations (88):
- China (88):
  - The First Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chao-yang Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Dong Zhi Men Hospital of Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Guang An Men Hospital China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - PLA Navy General Hospital, Beijing, Beijing Municipality
  - The Second Artillery General Hospital Of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Da Ping Hospital Of Third Military Medical University, Chongqing, Chongqing Municipality
  - Yongchuan Hospital Of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chinese People's Liberation Army No.180 Hospital, Quanzhou, Fujian
  - Chinese People's Liberation Army No.174 Hospital, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - 421 Hospital of PLA, Guangzhou, Guangdong
  - Guangdong Province Hospital of Traditional Chinese Medicine(TCM), Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi University of Chinese Medicine, Nanning, Guangxi
  - Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou
  - The Affiliated Baiyun Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital Of Zun Yi Medical College, Zunyi, Guizhou
  - Hainan Medical College Affiliated Hospital, Haikou, Hainan
  - Hainan Provincial Nong Ken Hospital, Haikou, Hainan
  - Affiliated Hospital of Cheng De Medical College, Chengde, Hebei
  - First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - Hebei Province Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei
  - TCM Hospital of Shi Jia Zhuang City, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Heilongjiang Provincial Academy of Traditional Chinese Medicine, Haerbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science And Technology, Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Huang Gang Central Hospital, Huanggang, Hubei
  - Hubei Provincial Hospital Of TCM, Wuhan, Hubei
  - Wuhan Integrated TCM & Western Medicine Hospital, Wuhan, Hubei
  - Zhong Nan Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiang Ya Hospital of Central South University, Changsha, Hunan
  - The Third Xiang Ya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Jiangsu Taizhou People's Hospital, Taizhou, Jiangsu
  - Taizhou Traditional Chinese Medicine Hospital, Taizhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Chinese People's Liberation Army No.94 Hospital, Nanchang, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Province People's Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital Of Jilin University, Changchun, Jilin
  - Dalian Municipal Central Hospital Affiliated Of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital Of Dalian Medical University, Dalian, Liaoning
  - First Affiliated Hospital of Liaoning Medical University, Jinzhou, Liaoning
  - People's Liberation Army No.202 Hospital, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Hospital Of China Medical University, Shenyang, Liaoning
  - The General Hospital Of Shenyang Military Region, Shenyang, Liaoning
  - Ningxia Hui Autonomous Region's Hospital, Yinchuan, Ningxia
  - The General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Jinan General Hospital of PLA, Jinan, Shandong
  - Qi Lu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Jining No.1 People's Hospital, Jining, Shandong
  - Chinese People's Liberation Army No.88 Hospital, Taian, Shandong
  - Yantai Yu Huang Ding Hospital, Yantai, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Chang Hai Hospital of the Second Military Medical University, Shanghai, Shanghai Municipality
  - Ren Ji Hospital of Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital Affiliated Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Xian, Shanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xian, Shanxi
  - Hua Xi Hospital of Sichuan University, Chengdu, Sichuan
  - First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Hospital of ITCWM, Nankai Hospital, Tianjin, Tianjin Municipality
  - The First Hospital of Shi He Zi Medical University, Shihezi, Xinjiang
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yan'an Hospital of Kunming City, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang L, Li P, Xing CY, Zhao JY, He YN, Wang JQ, Wu XF, Liu ZS, Zhang AP, Lin HL, Ding XQ, Yin AP, Yuan FH, Fu P, Hao L, Miao LN, Xie RJ, Wang R, Zhou CH, Guan GJ, Hu Z, Lin S, Chang M, Zhang M, He LQ, Mei CL, Wang L, Chen X. Efficacy and safety of Abelmoschus manihot for primary glomerular disease: a prospective, multicenter randomized controlled clinical trial. Am J Kidney Dis. 2014 Jul;64(1):57-65. doi: 10.1053/j.ajkd.2014.01.431. Epub 2014 Mar 14. PMID 24631042
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] Li P, Chen YZ, Lin HL, Ni ZH, Zhan YL, Wang R, Yang HT, Fang JA, Wang NS, Li WG, Sun XF, Chen XM. Abelmoschus manihot - a traditional Chinese medicine versus losartan potassium for treating IgA nephropathy: study protocol for a randomized controlled trial. Trials. 2017 Apr 11;18(1):170. doi: 10.1186/s13063-016-1774-6. PMID 28395659